CLINICAL TRIAL: NCT06518343
Title: The Trimethylamine N-oxide (TMAO)-Reducing Effects of a Pomegranate Supplement Simultaneously Administered With L-carnitine
Brief Title: Trimethylamine N-oxide Effects of a Pomegranate Supplement Simultaneously With Carnitine (TESSA)
Acronym: TESSA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: QIB01/2024; 336410 (Registry Identifier: IRAS)
Record Dates: First submitted 2024-07-19; First posted 2024-07-24 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2024-07

CONDITIONS: Healthy
MeSH Terms: interventions — Carnitine; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pomegranate extract (Experimental): 1.5 grams L-carnitine (Carnipure®) + 1.6 grams pomegranate extract (Dermogranate®) in hydroxypropyl methylcellulose (HPMC) capsules
  Interventions: Dietary Supplement: L-carnitine + Pomegranate extract
- Microcrystalline cellulose (Placebo Comparator): 1.5 grams L-carnitine (Carnipure®) + 1.5 grams microcrystalline cellulose (MCC, Redwells Health) in hydroxypropyl methylcellulose (HPMC) capsules
  Interventions: Dietary Supplement: L-carnitine + Microcrystalline cellulose

INTERVENTIONS:
Dietary Supplement: L-carnitine + Pomegranate extract — Participants will consume 1.5 grams L-carnitine with 1.6 grams pomegranate extract at one visit during one intervention period
  Arms: Pomegranate extract
Dietary Supplement: L-carnitine + Microcrystalline cellulose — Participants will consume 1.5 grams L-carnitine with 1.5 grams microcrystalline cellulose at one visit during one intervention period
  Arms: Microcrystalline cellulose

SUMMARY:
Trimethylamine N-oxide (TMAO) is produced in some individuals whose diets include meat, fish, and dairy.These foods are rich in L-carnitine. L-carnitine is metabolised by the liver and gut microorganisms (bacteria) into TMAO. In the TESSA study, investigators will explore whether pomegranate extract can lower the production of TMAO in healthy men and women. This reduction in TMAO production has been associated with decreasing a person's risk of heart disease.

DETAILED DESCRIPTION:
The TESSA study is a 18 day randomised, double-blind, placebo-controlled two-arm crossover pilot study conducted at the NIHR (National Institute for Health and Care Research) Norfolk Clinical Research Facility (CRF) in the Quadram Institute in Norwich. Investigators are seeking men and women over the age of 18 years who habitually consume meat, fish, and/or eggs and are TMAO producers to determine whether pomegranate extract affects L-carnitine metabolism compared to a matched placebo. This study is conducted in two phases. The first phase involves two study visits where investigators will identify and invite TMAO producing individuals to continue to the second phase of this study. Moreover, investigators will ask the participant to complete a food frequency questionnaire. The second phase involves two intervention periods which are separated by a 10 day washout. Each intervention period begins with a run-in followed by three study visits. Investigators will precisely quantify the absorption (blood plasma concentrations over time, pharmacokinetic study) and metabolism of L-carnitine and its products of metabolism which includes TMAO. Additionally, investigators will examine pomegranate metabolism and excretion with timed urine collections and stool samples.

Participants will consume three L-carnitine capsules at the first visit during the first phase. In the second phase, participants will consume L-carnitine capsules with the intervention capsules (pomegranate extract or placebo) for the first intervention period then after the washout period, participants will crossover and consume L-carnitine capsules with the other intervention capsules for the second intervention period. For each intervention period, three L-carnitine capsules with four intervention capsules at the first visit following the run-in. During the second phase starting at the run-in period participants will be asked to follow a standardized, controlled diet which will be low in choline, L-carnitine, and ellagitannins.

ELIGIBILITY:
Inclusion criteria (First phase):

* Individuals who regularly eat meat (4 portions of meat per week for at least 2 months prior to enrolment in the study).
* Aged 18 and older.
* Body Mass Index (BMI) between 18.5 - 30 kg/m2.
* Living within 40 miles from the Norwich Research Park.

Inclusion criteria (Second phase)

* meets first phase inclusion criteria
* TMAO producer (plasma TMAO increase of >5 µM and >50% after L-carnitine ingestion.

Exclusion criteria:

* Consume an entirely vegan, vegetarian, or pescatarian diet within the last two months.
* Do not have access to a freezer to store some provided meals and ice packs.
* Have a known allergy to the tablets, capsules (i.e., pomegranate), or standardised meals such as wheat, eggs, milk, nuts, and soybeans.
* Have difficulty swallowing, a swallowing disorder, or are unable to swallow four capsules (the size of a peanut) and three L carnitine tablets consecutively within a time span of ten minutes.
* Have bowel movements less than five times a week.
* Are a current smoker (or stopped smoking for less than 3 months).
* Consume more than 14 units of alcohol per week (for example, a pint of beer or a 175 mL glass of wine each count as two units).
* Are pregnant or breastfeeding.
* Have anaemia or any conditions or medications that may hinder clotting. This will be assessed on a case-by-case basis.
* Have high or low blood pressure (i.e., ≤90/60 or ≥160/100 mmHg).
* Have a medical condition or take medications that may affect the primary outcome of this study, such as but not limited to diabetes, liver disease, hypo/hyperthyroidism, or fish odour syndrome. This will be assessed on a case-by-case basis.
* Have had gastrointestinal disease or surgical procedures that may affect the primary outcome of this study. This will be assessed on a case-by-case basis.
* Have known or a history of kidney disease, this will be determined by the medical advisor using blood urea nitrogen and creatinine levels in the participant's blood.
* Regularly use bowel cleansing techniques like colonic irrigation or laxatives.
* Had an infection or received antibiotics within a month prior to this study.
* Regularly take dietary supplements that may affect the primary outcome measure of this study, such as fish oil or L carnitine supplements.
* Are currently undergoing active treatment for cancer or heart disease.
* Participated in another dietary intervention study within the last four months.
* Have donated a large quantity of blood within the last 16 weeks. Registered donors should abstain from blood donations for the duration of the study.
* Are a person related to or living with a member of the study team.
* Are unable to give written or verbal informed consent.
* Participant is unable to provide GP (General Practitioner) contact details.
* Have symptoms of Coronavirus infection (COVID-19), been asked to self-isolate, or have been diagnosed with COVID-19 in the last 14 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Difference in the area under the curve (AUC) of blood plasma TMAO concentrations after pomegranate extract and microcrystalline cellulose interventions. | Day 2,3,4,16,17,and 18
  Comparison of AUC of blood plasma TMAO concentrations after L-carnitine with pomegranate extract and after L-carnitine with microcrystalline cellulose interventions.

SECONDARY OUTCOMES:
Changes in area under the curve (AUC) from plasma concentrations of L-carnitine and its metabolites | 48 hours
  Plasma blood concentrations of L-carnitine and its metabolites (γ-BB: γ-butyrobetaine, TMA: trimethylamine, and TMAO) will be quantified after ingestion of L-carnitine and intervention capsules (pomegranate extract or microcrystalline cellulose). AUC will be determined using trapezoidal approximation of plasma concentrations over time. Measurements will be taken 0, 0.5, 1, 1.5, 2, 2.5, 16, 18, 20, 22, 24, and 48 hours after capsules have been ingested on Day 2 and Day 16.
Change in peak plasma concentration (Cmax) of L-carnitine and its metabolites | 48 hours
  Plasma blood concentrations of L-carnitine and its metabolites (γ-BB: γ-butyrobetaine, TMA: trimethylamine, and TMAO) will be quantified after ingestion of L-carnitine and intervention capsules (pomegranate extract or microcrystalline cellulose). Cmax will be the highest concentration measured during a 48 hour period. Measurements will be taken 0, 0.5, 1, 1.5, 2, 2.5, 16, 18, 20, 22, 24, and 48 hours after capsules have been ingested on Day 2 and Day 16.
Change in the time to reach peak plasma concentration (Tmax) of L-carnitine and its metabolites | 48 hours
  Plasma blood concentrations of L-carnitine and its metabolites (γ-BB: γ-butyrobetaine, TMA: trimethylamine, and TMAO) will be quantified after ingestion of L-carnitine and intervention capsules (pomegranate extract or microcrystalline cellulose). Tmax will be the time when peak concentration of L-carnitine or its metabolites has been reached. Measurements will be taken 0, 0.5, 1, 1.5, 2, 2.5, 16, 18, 20, 22, 24, and 48 hours after capsules have been ingested on Day 2 and Day 16.
Change in plasma half-life (t1/2) of L-carnitine and its metabolites | 48 hours
  Plasma blood concentrations of L-carnitine and its metabolites (γ-BB: γ-butyrobetaine, TMA: trimethylamine, and TMAO) will be quantified after ingestion of L-carnitine and intervention capsules (pomegranate extract or microcrystalline cellulose). Half life will be the time point where concentration of L-carnitine or its metabolites have reduced by half. Measurements will be taken 0, 0.5, 1, 1.5, 2, 2.5, 16, 18, 20, 22, 24, and 48 hours after capsules have been ingested on Day 2 and Day 16.
Change in the area under the curve (AUC) from urine concentrations of L-carnitine and its metabolites | 48 hours
  Urine concentrations of L-carnitine and its metabolites (γ-BB: γ-butyrobetaine, TMA: trimethylamine, and TMAO) will be quantified after ingestion of L-carnitine and intervention capsules (pomegranate extract or microcrystalline cellulose). AUC will be determined using trapezoidal approximation of plasma concentrations over time. Measurements will be taken from urine collections at 0, 2, 2.5 to 16, 18, 20, 22, 24, and 24 to 48 hours.
Change in pomegranate polyphenols and their metabolite concentrations from pooled 24 hour urine collections. | Day 3, 4, 17, and 18.
  Quantification of pomegranate polyphenols and their metabolite excretion into urine will be measured from pooled urine collections (24 and 48 hours) using targeted metabolite analysis of pomegranate polyphenols, punicalagin, ellagic acid, urolithins. These metabolites will be used to define relationships between dietary intake, pomegranate metabolism and pharmacokinetic outcomes
Difference in L-carnitine and its metabolites concentrations from faecal (stool) collections after pomegranate extract and microcrystalline cellulose interventions. | Day 2, 4, and 18.
  Comparison in L-carnitine and and its metabolite (γ-BB: γ-butyrobetaine, TMA: trimethylamine, and TMAO) excretion into faeces (stool) will be measured from faecal samples at baseline and after each intervention period. These metabolites will be used to define relationships between dietary intake, L-carnitine metabolism and microbiome composition
Changes in gut microbiota composition (indices of diversity and in taxonomic abundances) over study duration | Day 2, 4, 16, and 18.
  Comparison of gut microbiota composition will be determined using indices of diversity and taxonomic abundances using Shotgun metagenomic sequencing of faecal samples collected at the start and end of each intervention period.
Treatment effects of gut microbiota composition (indices of diversity and in taxonomic abundances) after pomegranate extract and microcrystalline cellulose interventions. | Day 4 and 18.
  Comparison of gut microbiota composition will be determined using indices of diversity and taxonomic abundances using Shotgun metagenomic sequencing of faecal samples collected at the end of each intervention period.
Difference in bacterial transcripts from faecal (stool) collections after pomegranate extract and microcrystalline cellulose interventions. | Day 2, 4, and 18.
  Comparison of absolute abundance of L-carnitine metabolising bacterial genes and their transcripts using specific qPCR (quantitative polymerase chain reaction) and RT-qPCR (Real-time polymerase chain reaction) assays from faecal samples collected at baseline and after each intervention period.
Correlation between plasma TMAO concentration and quantity of L carnitine-rich foods consumed in habitual diets of healthy men and women. | Phase 1 Day 2
  Plasma TMAO concentration measured during the first phase of this study will be correlated (Pearson correlation) with the quantity of L-carnitine-rich foods collected from a 90-day Food Frequency Questionnaire (VioCare VioScreen).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kroon, PhD, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Quadram Institute, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No